CLINICAL TRIAL: NCT05161000
Title: Effects of Oral Nutritional Supplementation With Dietary Counseling in Children at Risk of Undernutrition
Brief Title: Oral Nutritional Supplementation in Children at Risk of Undernutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AL48
Record Dates: First submitted 2021-12-03; First posted 2021-12-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Undernutrition
MeSH Terms: conditions — Malnutrition | interventions — Dietary Supplements; Nutrition Assessment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Nutritional Supplement (ONS) Group (Experimental): Two servings per day in addition to dietary counseling
  Interventions: Other: Oral Nutritional Supplement; Other: Dietary counseling
- Control Group (Other): dietary counseling
  Interventions: Other: Dietary counseling

INTERVENTIONS:
Other: Oral Nutritional Supplement — ONS plus dietary counseling
  Arms: Oral Nutritional Supplement (ONS) Group
Other: Dietary counseling — dietary counseling

SUMMARY:
The objective of this randomized, controlled trial is to evaluate the effects of consuming a pediatric oral nutritional supplement (ONS) plus dietary counseling for 120 days on anthropometric growth, strength, and nutritional status, compared with dietary counseling alone in undernourished children in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Child is 36 months - 107 months of age.
* Child is undernourished as determined by BMI for age z-score or Mid-upper-arm circumference z-score
* Child's caregiver has voluntarily signed and dated an informed consent form (ICF), approved by an IRB, and provided Health Insurance Portability and Accountability Act (HIPAA) or other applicable privacy regulation authorization prior to any participation in the study.
* Child's caregiver is willing to abstain from providing non-study oral nutrition supplements during the study period duration.
* Child's caregiver is able and willing to follow study procedures and record data in parent diaries and complete any forms or assessments needed during the study.
* Child is willing to consume the study product for the duration of the study, if randomized to intervention group

Exclusion Criteria:

* Child has a height-for-age z-score ≥ 0.
* Child is currently drinking an oral nutritional supplement (ONS) on a regular basis (≥ 15 days in the past month)
* Child is participating in another study that has not been approved as a concomitant study by AN.
* Child has been diagnosed with the following:

  * Galactosemia, or an allergy or intolerance to any ingredient found in the study product
  * Acute or chronic infections including but not restricted to respiratory infections, diarrhea, Hepatitis B or C, HIV infection or tuberculosis
  * Severe gastrointestinal disorders such as celiac disease, short bowel syndrome, pancreatic insufficiency, or cystic fibrosis
  * Neoplastic, renal, hepatic or cardiovascular, hormonal or metabolic disorders, Down's syndrome or significant, uncorrected cardiac anomalies that may impact growth
  * Infantile anorexia nervosa, developmental disability, including physical disorders such as cerebral palsy, or a developmental delay that is considered too severe for participation
  * Disorders of hemoglobin structure, function or synthesis
  * Clinically significant nutritional deficiency requiring specialty nutritional therapy
  * Any other clinically significant medical condition, which in the investigator's opinion, makes him or her unsuitable for inclusion in the study.

Ages: 36 Months to 107 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 279 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2024-06-11 (Actual)

PRIMARY OUTCOMES:
Weight-for-age z-score (WAZ) | baseline to 120 days
  Change in weight-for-age z-score

SECONDARY OUTCOMES:
Anthropometric Measurement Calculations | baseline to 120 days
  Standard z-scores and percentiles including weight-for-age, height-for-age, weight-for-height, BMI-for-age and mid-upper-arm-circumference-for-age
Mid-upper-arm circumference (MUAC) | baseline to 120 days
  Measured in cm
Weight | baseline to 120 days
  Measured in Kg
Height | baseline to 120 days
  Measured in cm
Dietary Diversity | baseline to 120 days
  Measured by 24-hour dietary recall
Appetite | baseline to 120 days
  Visual analog scale from Ate Very Little to Ate A Lot

OTHER OUTCOMES:
Hand Grip Strength | baseline to 120 days
  Measured in kg
Nutrition Biomarkers | baseline to 120 days
  Blood chemistry analysis of vitamin A, vitamin B12, vitamin D, vitamin E, folate, and vitamin K
Adverse Event Reporting | baseline to 120 days
  Standard adverse event reporting
Health Care Utilization | baseline to 120 days
  Number of unscheduled visits or missed school days (child) or work days (parent)
Sleep Data | baseline to 120 days
  Average daily number of hours
Activity Data | baseline to 120 days
  Average daily number of minutes
Physical Activity | baseline to 120 days
  Visual analog scale from Not Active to Very Active
Parental Stress Scale | baseline to 120 days
  18 questions scaled from Strongly disagree to Strongly Agree
Child Eating Behavior Questionnaire | baseline to 120 days
  35 questions 5-Point Likert Scale from Never to Always
Caregiver Opinion Questionnaire | baseline to 120 days
  3 Parent reported questions related to child's nutrition
Children's Sleep Habit Questionnaire | baseline to 120 days
  7 Parent reported questions related to child's sleep habits
Triceps Skinfold | baseline to 120 days
  Measured in mm

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Williams, MPH, Study Chair — Abbott Nutrition
Locations (17):
- United States (17):
  - Midway Medical Clinic, Oneonta, Alabama
  - HealthStar Research Glenwood, Glenwood, Arkansas
  - HealthStar Research, LLC, Hot Springs, Arkansas
  - L.A. Universal Research Center, Inc., Los Angeles, California
  - Kissimmee Clinical Research, Kissimmee, Florida
  - Dade Research Center, LLC, Miami, Florida
  - D&H National Research Centers, Miami, Florida
  - Suncoast Research, Assoc., LLC, Miami, Florida
  - Springs Medical Research, Owensboro, Kentucky
  - Velocity Clinical Research, Covington, Louisiana
  - Southern Clinical Research, Zachary, Louisiana
  - Alivation Research (Primary Care), Lincoln, Nebraska
  - Javara Inc. 3380, Winston-Salem, North Carolina
  - Tribe Clinical Research LLC., Greenville, South Carolina
  - Javara, Inc. 3377, Dallas, Texas
  - Proactive Clinical Research, Edinburg, Texas
  - Gentle Pediatrics, Sugar Land, Texas

IPD SHARING:
Plan to Share IPD: No